CLINICAL TRIAL: NCT07321041
Title: Effect of Neonatal Delivery Time on Umbilical Cord pH and Base Excess in Patients Undergoing Cesarean Section Under General and Spinal Anesthesia
Brief Title: Effect of Delivery Time on Umbilical Cord Blood Gas Parameters in Cesarean Sections Under General and Spinal Anesthesia
Acronym: DELTA-CS
Status: Not yet recruiting | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, murat sahin, Medical Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 4934
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Umbilical Cord Blood; Cesarean Section Surgery; General Anesthesia; Spinal Anesthesia; Blood Gas Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Anesthesia: This cohort includes pregnant women undergoing elective cesarean section under general anesthesia as part of routine clinical care. The anesthesia technique is selected based on standard clinical indications and patient preference, independent of study participation. No experimental intervention is applied. Neonatal delivery time and umbilical artery blood gas parameters (pH and base excess) are recorded prospectively for observational analysis.
- Spinal Anesthesia: This cohort includes pregnant women undergoing elective cesarean section under spinal anesthesia as part of routine clinical care. The anesthesia technique is determined according to standard clinical practice and patient preference, independent of study participation. No experimental intervention is performed. Neonatal delivery time and umbilical artery blood gas parameters (pH and base excess) are prospectively recorded for observational analysis.

SUMMARY:
The goal of this observational study is to evaluate the effect of neonatal delivery time on umbilical cord blood gas parameters in pregnant women undergoing elective cesarean section under general or spinal anesthesia. The study population consists of adult pregnant women aged 18-40 years with singleton term pregnancies scheduled for elective cesarean delivery.

The main questions it aims to answer are:

Is neonatal delivery time associated with changes in umbilical artery pH values under general and spinal anesthesia? Is neonatal delivery time associated with changes in umbilical artery base excess under general and spinal anesthesia? Researchers will compare cesarean sections performed under general anesthesia with those performed under spinal anesthesia to determine whether the relationship between delivery time and umbilical cord blood gas parameters differs between anesthesia techniques.

Participants will:

Undergo elective cesarean delivery under general or spinal anesthesia as part of routine clinical care Have neonatal delivery time recorded intraoperatively Have umbilical artery blood gas parameters (pH and base excess) measured immediately after birth as part of standard neonatal assessment

DETAILED DESCRIPTION:
This prospective, observational study will be conducted at a single tertiary care center and aims to investigate the relationship between neonatal delivery time and umbilical artery blood gas parameters in elective cesarean sections performed under general or spinal anesthesia. No experimental intervention will be applied, and all procedures will be carried out as part of routine clinical care.

Eligible participants will include adult pregnant women with singleton term pregnancies who are scheduled for elective cesarean delivery. The choice of anesthesia technique (general or spinal anesthesia) will be determined by standard clinical indications and patient preference, independent of study participation. No modification to anesthesia management or surgical technique will be made for the purposes of the study.

Neonatal delivery time will be defined as the interval between uterine incision and complete delivery of the neonate and will be recorded intraoperatively by the surgical team. Immediately after birth, umbilical artery blood samples will be obtained as part of routine neonatal assessment, and blood gas analysis will be performed to determine pH and base excess values.

Data will be collected using standardized case report forms and hospital electronic medical records. All data will be anonymized and coded prior to analysis to ensure participant confidentiality. The primary analyses will assess the association between neonatal delivery time and umbilical artery pH and base excess within each anesthesia group. Secondary analyses will compare blood gas parameters between general and spinal anesthesia groups after controlling for delivery time.

This study is expected to provide clinically relevant information regarding the impact of delivery time on neonatal metabolic status during cesarean delivery and to contribute to optimizing coordination between obstetric and anesthesia teams.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women aged 18-40 years Singleton pregnancy at ≥36+6 weeks of gestation Scheduled for elective cesarean section Planned delivery under general or spinal anesthesia Ability to provide written informed consent

-

Exclusion Criteria:

Emergency cesarean section Known fetal anomalies Multiple pregnancy Maternal comorbidities that may affect neonatal outcomes (e.g., diabetes mellitus, hypertension, preeclampsia) Conversion from spinal anesthesia to general anesthesia Failure to obtain umbilical artery blood gas sample or incomplete clinical data

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only female participants will be included, as the study population consists of pregnant women undergoing elective cesarean section.
Study Population: The study population consists of adult pregnant women aged 18-40 years with singleton term pregnancies who are scheduled for elective cesarean section under general or spinal anesthesia. All participants will be managed according to routine clinical practice, and no experimental intervention will be applied.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Umbilical Artery pH and Base Excess | Immediately after delivery
  Umbilical artery pH and base excess will be measured from arterial cord blood samples obtained immediately after delivery as part of routine neonatal assessment. These parameters will be used to evaluate neonatal metabolic status and their association with neonatal delivery time in cesarean sections performed under general and spinal anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Mus State Hospital, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as this is a single-center observational study using routinely collected clinical data. No predefined data-sharing agreement or repository is in place, and data sharing was not included in the original study protocol or ethics approval. De-identified aggregate results will be reported in publications.

REFERENCES:
- [Background] Kinoshita M, Sakai Y, Nakaji Y, Takahashi R, Matsumoto Y, Tanaka K. Factors influencing spinal anesthesia-to-delivery interval in elective cesarean sections: A retrospective analysis. Medicine (Baltimore). 2025 May 9;104(19):e42420. doi: 10.1097/MD.0000000000042420. PMID 40355198
- [Background] Hassanin AS, El-Shahawy HF, Hussain SH, Bahaa Eldin AM, Elhawary MM, Elbakery M, Elsafty MSE. Impact of interval between induction of spinal anesthesia to delivery on umbilical arterial cord ph of neonates delivered by elective cesarean section. BMC Pregnancy Childbirth. 2022 Mar 17;22(1):216. doi: 10.1186/s12884-022-04536-y. PMID 35300620